CLINICAL TRIAL: NCT04918316
Title: Initial Correction Keratoconus: Scleral vs Corneal Gas Permeable Lenses SCOPE Study
Brief Title: Initial Correction Keratoconus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Ellen S Shorter, Associate Professor of Clinical Ophthalmology, University of Illinois at Chicago
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2020-1504
Record Dates: First submitted 2021-05-14; First posted 2021-06-08 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Corneal gas permeable lens first (Active Comparator): Device: corneal gas permeable contact lenses (RoseK2 corneal Blanchard Contact Lens, Inc. Manchester, NH).
  Participants with an odd study ID will be fit with the corneal gas permeable lens first.
  Interventions: Other: Corneal gas permeable lens
- Scleral lens first (Active Comparator): Device: scleral lenses (SynergEyes VS (Synergeyes, Inc., Carlsbad CA).
  Participants with an even study ID will be fit with the scleral lens first.
  Interventions: Other: Corneal gas permeable lens

INTERVENTIONS:
Other: Corneal gas permeable lens — Fit in corneal gas permeable contact lens first.

SUMMARY:
Keratoconus is a non-inflammatory, progressive disease in which corneal irregularity increases. As the condition develops, more advanced forms of optical correction are needed to improve vision for patients. Until recently, small diameter corneal gas permeable lenses were considered the primary mode of correction for patients with keratoconus. Now, however, practitioners have multiple options for reducing the optical aberrations caused by keratoconus, including scleral lenses. As of yet, no single option for optical correction has been identified as the preferred mode of correction in terms of overall patient satisfaction with vision, comfort, and ease of use. The order in which various forms of optical correction would be most logically introduced has yet to be determined. This is a study comparing small diameter corneal gas permeable and large diameter scleral lenses in individuals with keratoconus.

This study will prospectively compare visual satisfaction and ease of use between corneal gas permeable and scleral lenses for patients with mild to moderate keratoconus.

DETAILED DESCRIPTION:
While both corneal gas permeable and scleral lenses have been show to improve visual acuity in individuals with keratoconus, it has yet to be determined if one option has superior comfort and overall patient satisfaction in patients new to gas permeable lens use. In this study, patients will be prospectively fit with both corneal gas permeable and scleral lenses according to standard clinical practice. Both corneal gas permeable and scleral lenses are considered standard of care for patients with keratoconus.

The investigators hypothesize that study participants will select scleral lens over corneal gas permeable lens as their preferred final lens type of choice.

The Primary outcome measure of this study is participant selected final lens choice for continued use for the management of keratoconus.

Methods:

Study Design This is a prospective, multi-center, randomized interventional clinical trial with a 2x2 crossover design of patients with keratoconus fit with corneal and scleral gas permeable contact lenses. The crossover design allows intra-subject differences between two randomized groups with participants serving as their own controls. Contact lens #1 will be the SynergEyes VS (Synergeyes, Inc., Carlsbad CA) which features bi-tangential toric peripheries with linear landing zones. The standard lens is 16.0mm and is available from 14.5 to 17.5mm diameters. Contact lens #2 will be the RoseK2 corneal gas permeable lens (Blanchard Contact Lens, Inc. Manchester, NH). The lens is available in with a base curve range from 4.30 to 8.60 mm, diameter of 7.90 to 10.40mm.

Inclusion Criteria

* Age 18 or older.
* Diagnosis of keratoconus.
* Available baseline corneal topography and pachymetry
* Amsler-Krumeich keratoconus classification of stage 1 or higher

Exclusion Criteria

* No prior corneal transplantation or INTACTS
* No prior use of hybrid, corneal or scleral gas permeable lenses
* Presence of corneal scarring

Study procedures During the initial study visits patient demographics, past ocular and medical history and best corrected visual acuity with manifest refraction will be recorded. Additional testing may include corneal topography, pachymetry and meibography. Dry eye symptoms and contact lens comfort will be assessed using the OSDI and CLDEQ questionnaires.

Participants will be fit according to standard practices with the RoseK 2 corneal gas permeable and Synergeyes VS scleral lenses following manufacturer's recommendations. Over refraction and best corrected visual acuity will be recorded. Subjective comfort with lens use rated on comfort scale of 0 (not comfortable) to 10 (very comfortable).

Participants will be randomized to dispense lens #1 vs lens #2. They will be trained in safe application and removal and provided instructions on lens disinfection procedures. Best corrected visual acuity with lens #1 and subjective comfort with lens use will be rated on comfort scale of 0 (not comfortable) to 10 (very comfortable).

At the next visit, participants will return wearing lens #1 for minimum of 3 hours. Best corrected visual acuity with lens #1 will be recorded as well as hours of lens wear today, average hours of lens wear time, days per week of per week and daily time spent on lens application and removal. They will rate subjective comfort with lens use on comfort scale of 0 (not comfortable) to 10 (very comfortable). Dry eye symptoms will be assessed using OSDI and CLDEQ questionnaires. Participants will be trained in application and removal with lens #2. Best corrected visual acuity with lens #2 and subjective comfort will be rated on comfort scale of 0 (not comfortable) to 10 (very comfortable).

At the final visit, participants will return wearing lens #2 for minimum of 3 hours. Best corrected visual acuity with lens #2 will be recorded as well as hours of lens wear today, average hours of lens wear time, days per week of per week and daily time spent on lens application and removal. They will rate subjective comfort with lens use on comfort scale of 0 (not comfortable) to 10 (very comfortable). Dry eye symptoms will be assessed using OSDI and CLDEQ questionnaires. Participants will be trained in application and removal with lens #2. Best corrected visual acuity with lens #2 and subjective comfort will be rated on comfort scale of 0 (not comfortable) to 10 (very comfortable).

The participant will make a final selection of lens of choice #1 or #2.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of keratoconus
* Available baseline corneal topography and pachymetry
* Amsler-Krumeich keratoconus classification9 of stage 1

Exclusion Criteria:

* No prior corneal transplantation or INTACTS
* No prior use of hybrid, corneal or scleral gas permeable lenses
* Presence of corneal scarring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Final contact lens choice | At study completion (6-24 weeks)
  Each study participant will select whether to continue with Lens 1 or Lens 2. The percentage of those who choose a Scleral Lens will be compared to the percentage of participants who select corneal gas permeable lenses.

SECONDARY OUTCOMES:
Subjective comfort with lens use | Baseline, Study Visit 1 (2-4 weeks), Study Visit 2 (4-10 weeks) and at study completion (6-24 weeks)
  Subjective comfort with lens use will be rated by participants on comfort scale of 0 (not comfortable) to 10 (very comfortable).

CONTACTS AND LOCATIONS:
Overall Officials: Ellen S Shorter, OD, Principal Investigator — University of Illinois at Chicago
Locations (4):
- United States (4):
  - University of Illinois at Chicago Eye and Ear Infirmary, Chicago, Illinois
  - Illinois Eye Institute, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - The Ohio State University College of Optometry, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT04918316/Prot_004.pdf
  • Informed Consent Form (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT04918316/ICF_005.pdf